CLINICAL TRIAL: NCT02019654
Title: An Investigation of the Biological and Neuronal Mechanisms of Post-Traumatic Stress Disorder, Depression and Post-Concussive Syndrome Onset Following a Traumatic Brain Injury
Brief Title: An Investigation of the Biological and Neuronal Mechanisms of Post Traumatic Stress Disorder, Depression and Post-Concussive Syndrome Onset Following a Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140032; 14-NR-0032
Record Dates: First submitted 2013-12-20; First posted 2013-12-24 (Estimated); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Traumatic Brain Injury; PTSD; Depression
Keywords: Post-Traumatic Stress Disorder (PTSD); Traumatic Brain Injury; Neuroendocrine; Epigenetics; Natural History
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Mild or moderate TBI within the past 30 days

SUMMARY:
Background: A traumatic brain injury (TBI) could mean a person is at high risk for other long-lasting problems. These problems could include post-traumatic stress disorder (PTSD), depression, and post-concussive syndrome (PCS). For example, about 700,000 Americans each year who have a TBI later go on to have PTSD also. Depression and PCS are also common in people who had a TBI. Some people will have these problems later. These problems can seriously interfere with a person s life. Some people will not have these problems at all. There are many reasons for this difference. Researchers think the main reason is that people have different genetic and environmental influences. Right now, we only have few kinds of treatments to prevent or treat these problems after a TBI. The few treatments we have often do not work well. It is important to understand what factors make a person at high risk for these problems after a TBI. This could allow researchers and doctors to help address these problems early. Addressing these problems earlier may help a person have better health in the long run.

Objectives:

* To study the biological changes that happen after mild to moderate TBI which could be linked to the onset of PTSD, depression, and post-concussive syndrome
* To study brain mechanisms that could explain risks for getting a psychiatric disorder after mild to moderate TBI. This will be done using a test called functional MRI (fMRI). This test takes images of the brain while a person is doing a simple task.

Eligibility:

* Men and women who are 18 to 65 years old.
* Had a mild to moderate TBI (including concussion) in the last month.

Design:

* 5 outpatient visits to the NIH Clinical Center over one year.
* The first visit is a screening visit to see if you can join the study. This visit must happen within 30 days of the TBI. The visit includes lab work (blood and urine), a history and physical exam done by a physician or nurse practitioner, and a psychiatric interview with a behavioral health nurse.
* Visits 2, 3, 4 and 5 happen at one, three, six and twelve months post-injury. At these visits participants may have some or all of the following tests: blood and saliva collection, urine collection, questionnaires and interviews to assess symptoms, a test to see your response to stress (called hydrocortisone challenge), and fMRI brain imaging.
* This study does not provide treatment.
* This study is not a substitute for seeing a primary care provider.
* This study should not replace any therapies you may be taking.

DETAILED DESCRIPTION:
Objective: A traumatic brain injury (TBI) places individuals at high risk for developing posttraumatic stress disorder (PTSD). TBIs account for the onset of PTSD in approximately 700,000 Americans each year. Depression and post-concussive syndrome (PCS) are also common and often comorbid with PTSD. However, even in this group, there is a high-level of inter-individual response to traumatic brain injuries, suggesting that a better understanding of the mechanisms underlying this risk would be of great value in directing preventive interventions. The reasons for this heterogeneity are undoubtedly multi-factorial, and involve a complex interplay between genetic and environmental factors, that we may be able to understand through peripheral biomarkers and central examination of neuronal functioning. We suggest that DNA methylation may be a putative biomarker of psychiatric risk, as it reflects long-term changes in the function of the gene and may shape the recovery ability of the TBI patient through changes in cell function. In addition, differential proteomic response, including the function of the neuroendocrine system, likely relates to changes from epigenetic modification in both neurons and immune cells, which may contribute to the risk for the onset of PTSD as well as depression and PCS. We have previously shown that both PTSD and depression are associated with endocrine alterations, leading us to question if this biological change may underlie vulnerability for the onset of PTSD as well as depression and PCS following a TBI. In support of the idea of shared vulnerability, patients with a TBI also often display endocrine function alterations. In addition, sleep disturbance is common following TBI and is a core symptom of PTSD depression and PCS, suggesting that sleep may contribute to psychiatric and neurological recovery from a TBI. This line of research is essential, as current treatments to prevent or treat psychiatric risk following TBI are often ineffective, and even treatment of PCS is limited. This poor understanding results in our limited ability to reduce the risk for compromises in the health and well-being of patients who sustain a TBI.

Study population: Participants with a moderate or mild TBI (n=100) will be followed for a period of one year.

Design: This is a natural history study that will recruit patients within 30 days of a mild/moderate TBI, and will follow them over a one year period, with follow-up at 1, 3, 6 and 12 months following the TBI. Biological profiles including the concentration of inflammatory proteins and neuropeptides, and DNA methylation will be examined. An optional structural and functional magnetic resonance imaging (fMRI), and a hydrocortisone stimulation test will be used to evaluate the role of neuronal and neuroendocrine functioning following TBI.

Outcome measures: The primary outcomes of interest are the biological changes that occur following TBI which are associated with the onset of psychiatric disorders of PTSD, and depression, as well as the onset of PCS. The secondary aim is to examine neuronal mechanisms that underlie the risks for these disorders through the use of fMRI. Additional aims will determine the role of psychological resilience traits in recovery and also how sleep relates to recovery and psychiatric risk.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must be enrolled in CNRM recruiting protocol (11-N-0084) or evaluated for a TBI at theGeorge Washington University Hospital, or referred from the NIH/CC Office of Patient Recruitment.
* Participants may be NIH employees/staff, except for those who are employed by NINR or subordinates, relatives, and/or co-workers of NINR employees/staff or study investigators.
* Participants will have had a mild to moderate TBI (GCS between 9 and 15) in the previous 30 days.
* Participants will be between the age of 18 and 65 years
* Ability to give own consent
* Demonstrate understanding of the protocol by passing a short consent quiz with a score of 6.

EXCLUSION CRITERIA:

* Psychiatric Risks: Actively suicidal or at risk for suicide
* Previous or current diagnosis of schizophrenia, bipolar disorder, other psychoses.
* Current diagnosis of depression.
* Previous or current PTSD.
* Current diagnosis of PCS.
* Current alcohol or drug abuse or dependence.
* Pregnancy.
* Under treatment for major illness or injury that may put the participant at higher risk during participation (such as: IV therapy for severe infections, chemotherapy for cancer, multiple necessary surgical interventions for injuries, unstable cardiac disease, severe immune dysfunction, etc.).
* History of any endocrine disorder or dysfunction, unless cleared via an endocrinology consult (including thyroid, adrenal and pituitary disorders).
* Abnormal lab values that may indicate endocrine disorder or dysfunction (unless cleared by endocrine consult) or that may suggest major illness as described above as determined by the screening clinician.
* Unstable diabetes.

Participant may be able to participate in the study but will not be able to have an MRI if they have any of the following:

* Metal in the body such as pacemakers, stimulators, pumps, aneurysm clips, metallic prostheses, artificial heart valves, cochlear implants or shrapnel fragments, or if they are a welder or metal worker.
* Claustrophobia
* Are not able to lie comfortably flat on their back for up to 90 minutes.

Participant may be able to participate in the MRI but not the Affective Stroop portion of the procedure if they are:

* Unable to see images close up without the aid of glasses (plastic goggles and contacts are permissible)
* Are unable to use their index and pointer fingers on both hands for the task.

Participants may not participate in the hydrocortisone stimulation testing if they have any of the following:

-History of any endocrine disorder or dysfunction, unless cleared via an endocrinology consult (including thyroid, adrenal and pituitary

disorders)

* Abnormal lab values that may indicate endocrine disorder or dysfunction (unless cleared by endocrine consult) or that may suggest major illness as described above as determined by the screening clinician.
* Diabetes Mellitus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will follow patients who sustained a mild or moderate TBI. Up to 120 participants (target n of completers = 100) will be enrolled into the study within 30 days of the TBI and will be followed over one year. Two groups will emerge: (1) those who develop PTSD, PCS, or depression and (2) those who are resistant to developing these disorders. Participants must be enrolled in CNRM recruiting protocol (11-N-0084), evaluated for a TBI at the George Washington University Hospital, or referred from the NIH/CC Office of Patient Recruitment. NIH employees may participate.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Examine proteomic concentrations of inflammatory proteins and neuropeptides following TBI and determine if these biomarkers relate to a greater risk for PTSD, depression or PCS. | Visit 1 (Month 1) and Visit 3 (Month 3)
  Protein concentrations of inflammatory proteins (IL-1, IL-6, CRP), and lower concentrations of neuropeptides (IGF-1, BDNF, galanin, NPY) and higher concentrations of (SB100, GFAP) collected at the first appointment will predict the onset of PTSD, depression or PCS.

SECONDARY OUTCOMES:
We will investigate the activation pattern and effective connectivity between the amygdala and other target regions regulating emotions (e.g., vmPFC or ACC) by analyzing fMRI data in patients following a TBI. We propose that the neurocircuitry-b... | Visits: 2, 3
  A model of neurocircuitry of acute stress onset based models of emotion regulation that emphasize the role of the amygdala and its reciprocal interactions with other target regions assessed through the use of a fMRI and the Affective Stroop Task.
Participants who develop PTSD, depression, or PCS will exhibit differential neuroendocrine functioning test responses using hydrocortisone stimulation test compared to controls who are resistant to these disorders. | Visits: 2,3,4,5
  A comparison of neuroendocrine functioning using the hydrocortisone stimulation between those cases that are compromised and develop PTSD, depression of PCS, and controls without these diagnoses.
Examine reported sleep quality following the TBI and determine if sleep disturbance is associated with the onset of PTSD, PCS or depression | Visits: 2,3,4,5
  The level of sleep disruption, as well as the reasons for disruption (i.e. sleep onset latency, frequent awakenings) between resistant and compromised participants. The relationship between self-reported health quality and symptomatology related to the development of PTSD, depression and PCS diagnoses.
Examine epigenetic modifications (i.e. DNA methylation) and genetic predisposition that may relate to the risk of developing PTSD, depression or PCS onset following a TBI. | Visits: 2,3,4,5
  Approximate multiple psychological constructs (i.e. fibromyalgia, chronic fatigue syndrome, etc), the relation between somatization and PTSD/TBI (and potentially the temporal order), and examine levels of overall somatization as a continuous variable across the entire cohort.
Compare the use of resilience traits/abilities in participants who develop PTSD, depression or PCS to TBI participants who are resistant to these disorders. | Visits: 2,3,4,5
  A profile of resilience abilities and traits that differ between resistant participants and compromised participants.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Camphausen, M.D., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-NR-0032.html